CLINICAL TRIAL: NCT03737864
Title: Native Center for Alcohol Research and Education (NCARE), Transition to Recovery
Brief Title: NCARE, Transition to Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 18-2421
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Withdrawal; Substance Use Disorders
Keywords: transition to substance abuse treatment; readmission; recidivism; patient navigation
MeSH Terms: conditions — Substance-Related Disorders; Recidivism | interventions — Patient Navigation; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview (Active Comparator): A single 45-60 minute 1:1 session of MI provided by patient navigators at discharged focused on transitioning patients to treatment after detoxification.
  Interventions: Behavioral: Motivational interviewing (MI)
- Patient navigation and MI (Experimental): A single 45-60 minute 1:1 session of MI provided by patient navigators at discharged focused on transitioning patients to treatment after detoxification plus patient navigation for 30 days, or until the patient is successfully enrolled in substance abuse treatment, or readmission to detoxification occurs, whichever occurs first.
  Interventions: Behavioral: Patient navigation

INTERVENTIONS:
Behavioral: Patient navigation — The patient navigator will provide support to patients upon discharge and will maintain regular contact either in person or by phone at a minimum of once per week for 30 days, or until the patient successfully enrolled in substance abuse treatment, or readmission to detoxification occurs, whichever occurs first.
  Arms: Patient navigation and MI
Behavioral: Motivational interviewing (MI) — A single 45-60 minute 1:1 session of MI provided by patient navigators at discharged focused on transitioning patients to treatment after detoxification.
  Arms: Motivational Interview

SUMMARY:
This study tests the effectiveness of patient navigation for increasing enrollment in substance abuse treatment programs and preventing readmission to detoxification. Participants will be randomized to receive motivational interviewing or motivation interviewing plus patient navigation.

DETAILED DESCRIPTION:
The primary goal of alcohol detoxification is to medically manage acute intoxication and withdrawal. Its secondary goal of fostering entry into longer-term alcohol treatment post-detoxification is often overlooked. This leads to a revolving door characterized by a cyclical pattern of discharges and re-admissions to detoxification. This pattern is observed across the US among alcohol detoxification patients and is even more prevalent among Alaska Native people; few transition to alcohol treatment following detoxification and approximately 40% are readmitted within 1 year. The revolving door is costly to patients and providers. Current estimates associated with the cost of detoxification are not available. A study over 25 years ago indicated the average inpatient detoxification stay was over $3,300. Although the Substance Abuse and Mental Health Administration recognizes that better linkages are needed to transition people to treatment following detoxification, few interventions have tested ways to improve this transition; none of these prior studies included either Alaska Natives or American Indians.

This study proposes to use patient navigators to guide and assist patients in their transition to the appropriate levels of treatment, and to help eliminate barriers that obstruct treatment entry. This is a randomized controlled trial of the patient navigation intervention with 612 patients. We will estimate the costs of implementing and sustaining this intervention as well as its economic value. The control condition will include 1 session of motivational interviewing lasting approximately 45 minutes to 1 hour. The intervention group will also receive motivational interviewing and in addition will work with a patient navigator to facilitate entry into the appropriate level of care and provide ongoing support until the patient is admitted to treatment or the intervention period ends.

Specific Aims:

1. Adapt patient navigation (Transitions to Recovery) to fit the patient population and test its effectiveness in increasing successful transition to post-detoxification substance abuse treatment.
2. Test patient navigation's effectiveness in preventing readmission to detoxification.
3. Perform a comprehensive economic evaluation of patient navigation (Transition to Recovery) by using cost-benefit analyses.

If effective, this intervention may be a cost-effective means of transitioning detoxification patients to treatment across health care systems nationally.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* successful completion of the detoxification process (completion of the detoxification process is a necessary step in order to transitions to substance abuse treatment) from our partnering detoxification facility.
* no comorbid physical or mental health condition (e.g., cancer, severe suicidality) that would delay transition to alcohol treatment.
* willing and cognitively able to provide informed consent and complete all study procedures assessed by detoxification discharge nurses.
* not currently admitted to a substance abuse treatment program

Exclusion:

* discharge destination prison or jail
* already enrolled in substance abuse treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Transition to substance abuse treatment | 30 days
  The date of entry into a substance abuse treatment program will be collected. A calculated a variable that reflects the number of days between detoxification discharge and transition to substance abuse treatment, and a binary indicator of successful transition to treatment within 0 to 30 days.

SECONDARY OUTCOMES:
Readmission to detoxification | 1 year
  Extract the date of the first readmission (if one occurs) or collect at 6 and 12 month follow-up following discharge from detoxification and calculate a variable indicating total days to readmission within one year.

CONTACTS AND LOCATIONS:
Overall Officials: Spero M Manson, PhD, Principal Investigator — University of Colorado, Denver; Michael McDonell, PhD, Study Director — Washington State University
Locations (1):
- Gateway to Recovery, Fairbanks, Alaska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Running Bear U, Poole EM, Muller C, Hanson JD, Noonan C, Trojan J, Rosenman R, Manson SM. The use of patient navigation to transition detoxification patients to substance use treatment in the Alaska Interior. Public Health Pract (Oxf). 2023 Aug 6;6:100418. doi: 10.1016/j.puhip.2023.100418. eCollection 2023 Dec. PMID 37635913